CLINICAL TRIAL: NCT02493062
Title: Evaluation of Hysterotomy Site After Open Fetal Surgery
Acronym: Hysterotomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment below the target goal; statistical analysis unable to be completed.
Sponsor: St. Louis University (Other)
Collaborators: SSM Health (Other)
Responsible Party: Principal Investigator, Laura Vricella, MD, MD, FACOG, Assistant Professor, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FCI-22581
Record Dates: First submitted 2015-06-03; First posted 2015-07-09 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Myelomeningocele; Pregnancy
Keywords: Hysterotomy; Myelomeningocele; Open fetal surgery; Sonohysterogram
MeSH Terms: conditions — Meningomyelocele | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single-arm study (Experimental): This single-arm study is described by women who have undergone prenatal fetal open (uterus was opened to perform a fetal intervention/surgery) surgery and cesarean section delivery. These women will undergo sonohysterogram.
  Interventions: Device: Sonohysterogram

INTERVENTIONS:
Device: Sonohysterogram — The sonohysterogram can measure the size and depth of the uterine scar allowing better predictive values for future pregnancies.
  Other Names: ultrasound

SUMMARY:
This study is to review how the uterus heals after having open fetal surgery. Open fetal surgery causes a scar perhaps two: one from the open fetal surgery and a second from delivery by cesarean section; rarely, the same area of your uterus was used for both open fetal surgery and delivery. From other studies of surgery performed on a uterus, some of the uterine scars do not heal well. This study's intervention uses sterile saline to spread open the inside of the uterus. The saline is slowly injected into the uterus using a catheter. An ultrasound called a sonohysterogram is performed to take pictures of the uterus, its inside and the walls of the uterus. In this way, the healed areas from the uterine surgery can be seen with ultrasound and evaluated. This is performed at least 6 months after delivery.

Primary Outcome:

Measure the depth of the scar and location of the scar 6 months or longer after delivery.

DETAILED DESCRIPTION:
This is an Investigator initiated, prospective study reviewing medical records and performing a sonohysterogram on non-pregnant women at 6 or more months after delivery of an infant who received open fetal repair.

An evaluation is completed at SSM Cardinal Glennon (CG), Fetal Care Institute (FCI) of a woman who has decided to have open fetal surgery to complete a fetal repair before the infant is born.

* After open fetal surgery participant will be monitored and delivered appropriately.
* After the infant is born investigators will review the mother's and infant's electronic health records and FCI database records
* 6 months or more after delivery of an infant who has received open fetal repair the participant will go to Saint Louis University (SLU) Care for a sonohysterogram to evaluate the healing process.

ELIGIBILITY:
Inclusion Criteria:

* SSM Cardinal Glennon Fetal Care Institute evaluation
* Received Open Fetal Surgery
* Open fetal surgery of myelomeningocele: maternal age of >= 18 yrs. and <=50 yrs.
* If a woman < 18 years old presented with a fetal tumor requiring open fetal repair, this would be done if deemed ethically sound by both CG and St. Mary's Health Center (SMHC) ethics committees. Given this, then the patient may qualify for this study. This is a RARE event.
* Agree to travel to SSM St. Mary's in St. Louis for sonohysterogram 6 or more months after delivery.

Exclusion Criteria:

* Presently pregnant
* Hysterectomy after delivery
* Menopause
* Using IUD (Intrauterine Device) for birth control
* There is no exclusion criteria for infants

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-06; Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vricella, MD, Principal Investigator — St. Louis University
Locations (1):
- SSM Cardinal Glennon Fetal Care Institute, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Enrollment was below the target enrollment goals therefore statistical analysis was not completed.

REFERENCES:
- See also: SSM Cardinal Glennon Fetal Care Institute Website — https://www.ssmhealth.com/cardinal-glennon/fetal-care-institute

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was June, 2013 through August, 2016. Patients were recruited for study during fetal surgery evaluation in the St. Louis Fetal Care Institute office. If patients were interested in participating in the study, the research nurse contacted the patient after delivery and set up an appointment at 6 months postpartum.
Groups:
- Single-arm Study: This single-arm study is described by women who have undergone prenatal fetal open (uterus was opened to perform a fetal intervention/surgery) surgery and cesarean section delivery.
  Sonohysterogram: The sonohysterogram can measure the size and depth of the uterine scar allowing better predictive values for future pregnancies.
Period: Overall Study
Arm/Group | Single-arm Study
Started | 35
Completed | 23
Not Completed | 12
Not completed — Physician Decision | 12

BASELINE CHARACTERISTICS:
Population: The baseline participants are the women that completed the study.
Arm/Group | Single-arm Study
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 28 [20 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Cesarean Hysterotomy Myometrial Thickness
Description: Average myometrium thickness surrounding niche is measured by measuring Average thickness of the myometrium toward the cervix and toward the fundus resulting in the average myometrium thickness surrounding the niche, measured by the sonohysterogram.
Time Frame: Minimum of 6 months after delivery.
Measure: Mean (Full Range); unit: millimeter
Arm/Group | Single-arm Study
Number analyzed (Participants) | 23
millimeter | 1.11 [0.56 to 1.68]

2. Primary Outcome: Cesarean Hysterotomy Site Myometrial Percentage of Thinning at the Niche
Description: Average myometrium will be calculated, measured by the sonohysterogram. The myometrium will be measured caudad and cephalad of the niche and averaged ((Caudad side in mm + Cephalad side in mm)/2)=Average myometrium thickness The myometrium at niche will be measured (niche mm). Average myometrium-niche mm= niche thinning (mm).
  Niche thinning / Average myometrium thickness= Percentage of thinning at the niche.
  Ex:
  Average thickness at niche: 0.5 mm Caudad myometrium thickness: 1.5 mm Cephalad myometrium thickness: 1.5 mm
  1.5mm + 1.5mm= 3mm/ 2= 1.5mm (average Myometrium Thickness)
  1.5mm- 0.5mm = 1.0 mm (Niche thinning)
  0.5mm / 1.0 mm (% of thinning at the niche)
Time Frame: Minimum of 6 months after delivery.
Measure: Mean (Full Range); unit: percentage of thinning
Arm/Group | Single-arm Study
Number analyzed (Participants) | 23
percentage of thinning | 44 [0 to 85]

3. Primary Outcome: Fetal Myelomeningocele Hysterotomy Site Myometrial Thickness
Description: Average myometrium thickness surrounding niche is measured by measuring average thickness of the myometrium to the right and left of the niche resulting in the average myometrium thickness surrounding the niche. This is measured by the sonohysterogram.
Time Frame: Minimum of 6 months after delivery.
Measure: Median (Full Range); unit: millimeter
Arm/Group | Single-arm Study
Number analyzed (Participants) | 23
millimeter | 1.37 [0.91 to 2.08]

4. Primary Outcome: Fetal Myelomeningocele Hysterotomy Site Myometrial Percentage of Thinning at the Niche
Description: Average myometrium will be calculated, measured by the sonohysterogram. The myometrium will be measure to the right and left of the niche and averaged ((Right side in mm + Left side in mm)/2)=Average myometrium thickness The myometrium at niche will be measured (niche mm). Average myometrium-niche mm= niche thinning (mm).
  Niche thinning / Average myometrium thickness= Percentage of thinning at the niche.
  Ex:
  Average thickness at niche: 0.5 mm Right sided myometrium thickness: 1.5 mm Left sided myometrium thickness: 1.5 mm
  1.5mm + 1.5mm= 3mm/ 2= 1.5mm (average Myometrium Thickness)
  1.5mm- 0.5mm = 1.0 mm (Niche thinning)
  0.5mm / 1.0 mm (% of thinning at the niche)
Time Frame: Minimum of 6 months after delivery.
Measure: Mean (Full Range); unit: percentage of thinning at the niche
Arm/Group | Single-arm Study
Number analyzed (Participants) | 23
percentage of thinning at the niche | 33 [12 to 73]

5. Primary Outcome: Percent of Participants With/Without Dehiscence (>80% Thinning of the Myometrium) at the Niche
Description: Yes >80% of thinning of the myometrium at the niche or No < 80% of thinning of the myometrium at the niche of the hysterotomy measured by the sonohysterogram.
Time Frame: Minimum of 6 months after delivery.
Measure: Number; unit: percentage of patients with >80% thinnin
Arm/Group | Single-arm Study
Number analyzed (Participants) | 23
percentage of patients with >80% thinnin
  Dehisence | 0
  No Dehisence | 100

ADVERSE EVENTS:
Time Frame: The study was conducted at 6 months or longer after delivery. The shortest time period was 6 months and the longest time period was 2 years from the date of delivery.
Arm/Group | Single-arm Study
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

LIMITATIONS AND CAVEATS:
Enrollment was below the target enrollment goals therefore statistical analysis was not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT02493062/Prot_SAP_000.pdf